CLINICAL TRIAL: NCT06301633
Title: Comparison of Oral and Nasal Tube Feeding on Stroke-related Dysphagia: A Prospective Multicenter Study
Brief Title: Comparison of Oral and Nasal Tube Feeding on Stroke-related Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOE-STROKE
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oro-esophageal Tube Feeding+comprehensive rehabilitation therapy (Experimental): Study lasts 15 days for each patient. The patients were given comprehensive rehabilitation therapy. The observation group was provided the support of enteral nutrition by Intermittent Oro-esophageal Tube Feeding.
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: comprehensive rehabilitation therapy
- Nasogastric Tube Feeding+comprehensive rehabilitation therapy (Active Comparator): Study lasts 15 days for each patient. The patients were given comprehensive rehabilitation. The observation group was provided the support of enteral nutrition by Nasogastric Tube Feeding.
  Interventions: Device: Nasogastric Tube Feeding; Behavioral: comprehensive rehabilitation therapy

INTERVENTIONS:
Device: Intermittent Oro-esophageal Tube Feeding — The specific procedure was as follows: the infant was placed in a semi-recumbent or sitting position with the head fixed. Before each feeding, the infant's oral and nasal secretions were to be cleared. An intermittent oro-esophageal tube was appropriately lubricated with water on the head part. The professional medical staff held the tube and slowly inserted it through one side of the mouth into the upper part of the esophagus. The depth of insertion depended on the patient's age and height. After each feeding, the tube was immediately removed, and the patient was held upright for at least 30 minutes in case of reflux.
  Arms: Intermittent Oro-esophageal Tube Feeding+comprehensive rehabilitation therapy
Device: Nasogastric Tube Feeding — Nasogastric Tube Feeding were used for feeding to provide nutritional support. Each feeding was administered by a nurse using the infant's mother's breast milk through the tube. The amount of each feeding varied from 20 to 100 ml depending on the age of the infant, with feedings given every 2 to 3 hours, approximately 10 times per day. The duration of each feeding procedure ranged from 10 to 20 minutes. The total daily intake ranged from 200 to 1000 ml. Each tube was kept indwelling for 5 to 7 days. When the tube needed to be replaced, it was removed after the last feeding of a day and a new tube was to be inserted through the other nostril on the following morning to continue the nutritional support.
  Arms: Nasogastric Tube Feeding+comprehensive rehabilitation therapy
Behavioral: comprehensive rehabilitation therapy — Both groups were given comprehensive rehabilitation therapy. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.

SUMMARY:
This was a prospective multicenter study. the patients after stroke with were randomly divided into the observation group and the control group. All patients were given comprehensive rehabilitation therapy. During the treatment, enteral nutrition support was provided for the two groups by Intermittent Oro-esophageal tube feeding and nasogastric tube feeding, respectively. Nutritional status, dysphagia, quality of life and depression before and after treatment were compared.

DETAILED DESCRIPTION:
Dysphagia in patients after stroke continues to be a challenge. To avoid the wound caused by gastrostomy, nasogastric tube feeding has been the mainstay of palliation, but potential side effects exist this choice. Intermittent Oro-esophageal tube feeding is an established modality that can be used with comprehensive rehabilitation therapy. This study reports the outcomes of Intermittent Oro-esophageal tube feeding and comparison with nasogastric tube feeding, including nutritional status, dysphagia, quality of life, depression, and follow-up in patients receiving comprehensive rehabilitation therapy.This was a prospective multicenter study. the patients after stroke with were randomly divided into the observation group and the control group. All patients were given comprehensive rehabilitation therapy. During the treatment, enteral nutrition support was provided for the two groups by Intermittent Oro-esophageal tube feeding and nasogastric tube feeding, respectively. Nutritional status, dysphagia, quality of life and depression before and after treatment were compared.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* meeting the diagnostic criteria of stroke;
* any degree of dysphagia at admission;
* steady vital signs, without severe cognitive impairment or sensory aphasia, able to cooperate with the assessment.
* transferred out within three weeks of hospitalization in the neurology department.

Exclusion Criteria:

* complicated with other neurological diseases;
* damaged mucosa or incomplete structure in nasopharynx;
* tracheostomy tube plugged;
* unfeasible to the support of parenteral nutrition;
* simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 15
  Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. The scores ranged 1 point to 8 points. As the level increased, the severity of dysphagia also increased.

SECONDARY OUTCOMES:
Body weight | day 1 and day 15
  Body weight measurement of the infants was conducted by the same nurse according to the relevant standards.
total protein | day 1 and day 15
  The relevant indicators include total protein (TP, g/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach infants and in the morning.
albumin | day 1 and day 15
  The relevant indicators include albumin (ALB, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach infants and in the morning.
Yale pharyngeal residue severity rating scale | day 1 and day 15
  The Yale pharyngeal residue severity rating scale was recruited for assessment, of which the result would be divided into 5 levels (1, no residue; 2, the covered pharyngeal mucosa; 3, mild residue, less than 50%; 4, moderate residue, more than 50%; 5, severe residue, spillage from laryngeal vestibule observed).As the level increased, the severity of dysphagia also increased.
Patient health questionnaire-9 | day 1 and day 15
  The depression of the patients was evaluated with the patient health questionnaire-9. The scores ranged 0-27. As the scores increased, the severity of depression also increased.
Swallowing Quality of Life questionnaire | day 1 and day 15
  Swallowing Quality of Life questionnaire was used to evaluate the quality of life, which consists of 44 items and divided into 11 main domains, including: overall satisfaction, understanding, diet, hydration, communication, respiratory issues, postoperative recovery, social impact, mental health, saliva control, and appearance. The maximum rough score was 220 points, which was converted into a standard percentage system in our study. As the scores increased, the quality of life was better.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group
Locations (1):
- The 1st afi. Hos., Zhenzhou, China

IPD SHARING:
Plan to Share IPD: No